CLINICAL TRIAL: NCT01686113
Title: Free Fatty Acids: Short Exposure Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Purdue University (Other)
Responsible Party: Principal Investigator, Richard Mattes, Distinguished Prof Foods and Nutrition, Purdue University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 1205012317
Record Dates: First submitted 2012-09-12; First posted 2012-09-17 (Estimated); Last update posted 2014-11-21 (Estimated); Status verified 2014-11

CONDITIONS: Hypogeusia
Keywords: Taste; Fat Taste; Threshold Testing
MeSH Terms: conditions — Ageusia | interventions — Fatty Acids, Nonesterified; Oleic Acid; Sucrose

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- NEFA (Experimental): Participants swish and spit 5 mL of an oleic acid solution everyday for 10 days.
  Interventions: Other: NEFA
- Control (Active Comparator): Participants swish and spit 5 mL of sucrose solution everyday for 10 days.
  Interventions: Other: Sucrose

INTERVENTIONS:
Other: NEFA
  Other Names: Oleic acid
  Arms: NEFA
Other: Sucrose
  Arms: Control

SUMMARY:
This study will examine whether or not short, daily exposures change a person's ability to detect free fatty acids in a solution by its taste. Repeated exposure should improve a person's ability to detect free fatty acids.

DETAILED DESCRIPTION:
The possibility that humans can taste non-esterified fatty acids (NEFA) - so-called fat taste - is a relatively new area of research. Previous work suggests that subjects require an average of between two and three testing sessions of approximately an hour each before they can reliably detect NEFA, and the average number of visits to get the lowest threshold is six. Streamlining this process is of great interest to researchers who wish to test many people as quickly as possible. Other taste qualities, including umami and sweet, have shown improvement in detection sensitivity in subjects that have undergone ten second exposures to these taste qualities for 10 days upon subsequent re-testing. We seek to determine if the same improvements can be seen with fat taste.

ELIGIBILITY:
Inclusion Criteria:

* good health
* available for multiple testing visits

Exclusion Criteria:

* have participated in a fat taste study in the past 6 months

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2012-05; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
NEFA detection threshold | 10 days

SECONDARY OUTCOMES:
Hunger | 2 days
  Visual analog scale assessment of hunger level prior to testing
BMI | 1 day
Taste descriptor | 10 days
  Description of NEFA taste by participant, e.g., sour, bitter, etc.

CONTACTS AND LOCATIONS:
Overall Officials: Richard D Mattes, PhD, Principal Investigator — Purdue University
Locations (1):
- Purdue University, West Lafayette, Indiana, United States